CLINICAL TRIAL: NCT01734525
Title: A Pilot Study for the Use of Biomarkers and Early Treatment of Invasive Candidiasis in ICU Patients
Brief Title: Negative Beta Glucan in ICU Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Marcio Nucci, MD, Universidade Federal do Rio de Janeiro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Early Therapy
Record Dates: First submitted 2012-11-20; First posted 2012-11-27 (Estimated); Results first posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-04

CONDITIONS: Candidemia
Keywords: candidemia; intensive care unit; 1,3 beta-D-glucan
MeSH Terms: conditions — Candidemia | interventions — Anidulafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anidulafungin (Experimental): Patients at risk will receive therapy with anidulafungin
  Interventions: Drug: Anidulafungin

INTERVENTIONS:
Drug: Anidulafungin — Anidulafungin at a dose of 200 mg in the first day and 100 mg daily afterwards

SUMMARY:
This is a prospective study aimed at testing a strategy of early initiation of an antifungal agent to patients admitted to intensive care units (ICUs) at risk for invasive candidiasis. Score system have been developed to identify groups at very high risk for the development of candidemia/invasive candidiasis in the ICU. These scoring system have used clinical information with or without data on Candida colonization, and have shown reasonable correlation with candidemia/invasive candidiasis. More recently, a biomarker - detection of 1,3-beta-D-glucan in the serum - has been tested in the early diagnosis of candidiasis. The incorporation of biomarkers such as beta-D-glucan could help clinicians to select a group at higher risk for candidemia, and despite the fact that these tests may give false-positive results, their negative predictive value could be of great help.

Therefore, the objectives of this study are:

1. To assess the frequency of positive biomarkers in ICU patients at high risk to develop invasive candidiasis/candidemia;
2. To test the strategy of early discontinuation of antifungal therapy based on repeatedly negative blood cultures and 1,3 beta-D-glucan in the serum.

DETAILED DESCRIPTION:
Entry criteria are: In the ICU for >2 days AND systemic antibiotics >2 days OR central venous catheter for >days AND at least two of the following: total parenteral nutrition, dialysis, surgery, pancreatitis, receipt of corticosteroids, receipt of other immunosuppressive agents. In addition, patients must have a clinical sign of infection (either one of the following): fever, hypothermia, hypotension, unexplained acidosis, or unexplained elevation in C-reactive protein.

Eligible patients will be enrolled after signing an informed consent and will have blood obtained for culture and determination of 1,3 beta-D-glucan serum levels for 3 days, and will start anidulafungin IV.

If all tests are negative, anidulafungin will be discontinued on day 4. If 1,3 beta-D-glucan is positive (>80 pg/ml) and / or blood cultures are positive for Candida species, anidulafungin will be continued for >14 days.

ELIGIBILITY:
Inclusion Criteria:

* In the ICU for >2 days AND

  * Systemic antibiotics on days 1-3 of ICU OR
  * Central venous catheter on days 1-3 of ICU
* AND at least 2 of:

  * Total parenteral nutrition on days 1-3 of ICU
  * Any dialysis on days 1-3 of ICU
  * Major surgery in the 7 days before admission in the ICU
  * Pancreatitis in the 7 days before admission in the ICU
  * Use of corticosteroids for at least 3 days in the 7 days before admission
  * Use of other immunosuppressive agents in the 7 days before admission in the ICU
* In addition, the patient must have at least one of the following:

  * Fever (axillary temperature >37.5 oC)
  * Hypothermia (axillary temperature <35 oC)
  * Hypotension
  * Unexplained acidosis
  * Unexplained elevation in C-reactive protein

Exclusion Criteria:

* Antifungal for >3 days
* Allergy to an echinocandin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcio Nucci, MD, Study Chair — Universidade Federal do Rio de Janeiro
Locations (1):
- Federal University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Nucci M, Nouer SA, Esteves P, Guimaraes T, Breda G, de Miranda BG, Queiroz-Telles F, Colombo AL. Discontinuation of empirical antifungal therapy in ICU patients using 1,3-beta-d-glucan. J Antimicrob Chemother. 2016 Sep;71(9):2628-33. doi: 10.1093/jac/dkw188. Epub 2016 Jun 10. PMID 27287231

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anidulafungin
Started | 85
Completed | 85
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Anidulafungin
Number analyzed (Participants) | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 40
Age, Continuous [Median (Full Range); unit: years] | 63 [22 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 41
Region of Enrollment [Number; unit: participants]
  Brazil | 85

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Ocurrence of Candidemia in Patients With Negative 1,3 Beta-D-glucan Who Discontinue Anidulafungin
Description: The main interest is to evaluate the ocurrence of candidemia in patients with negative 1,3 beta-D-glucan who discontinue anidulafungin
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 21
Participants
  Candidemia | 0
  No candidemia | 21

ADVERSE EVENTS:
Groups:
- One Arm: Patients at risk will receive therapy with anidulafungin
  Anidulafungin: Anidulafungin at a dose of 200 mg in the first day and 100 mg daily afterwards
Arm/Group | One Arm
Serious Adverse Events (participants affected / at risk) | 0/85
Other Adverse Events (participants affected / at risk) | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No